CLINICAL TRIAL: NCT02905422
Title: Healthy Eating, Activity, & Lifestyle Training Headquarters: II (H.E.A.L.T.H -II) Pilot Project
Brief Title: Healthy Eating, Activity, & Lifestyle Training Headquarters: II Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Tiffany Stewart, Associate Professor, Director, Behavior Technology Laboratory, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PBRC 2015-013
Record Dates: First submitted 2016-09-07; First posted 2016-09-19 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Overweight; Weight Loss
Keywords: physical activity; sleep; nutrition; Soldier; prevention; remote monitoring; mobile technology
MeSH Terms: conditions — Overweight; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist Control Group (No Intervention): Six month delayed access to the H.E.A.L.T.H. II Intervention - Intensive intervention (wait-list control)
- Active Intervention Group (Active Comparator): Immediate access to the H.E.A.L.T.H. II Intervention - Intensive intervention
  Interventions: Behavioral: H.E.A.L.T.H. II Intervention

INTERVENTIONS:
Behavioral: H.E.A.L.T.H. II Intervention — 12 month study with 6 month intervention phase and 6 month follow up phase. Participants will receive bi-weekly educational information pertaining to weight loss during the intervention phase. Participants will use online website to monitor weight, access meal plans, access weight loss information, and access fitness plans.
  Other Names: Army H.E.A.L.T.H. Intensive
  Arms: Active Intervention Group

SUMMARY:
The proposed study aims to combine evidenced based tools and guidance (H.E.A.L.T.H.: Healthy Eating Activity Lifestyle Training Headquarters) previously tested that has been developed specifically for use by Army Soldiers and a remote clinical intervention model that includes mobile tracking technology/devices for physical activity, weight and nutrition. This program is called the H.E.A.L.T.H. Intensive.

DETAILED DESCRIPTION:
The purpose of this investigation is to test the efficacy of a remote intervention to assist Soldiers in meeting standards for body fat and fitness. The intervention will include:

1. An Internet/Smartphone program for weight management and weight gain prevention developed during previous DoD research.
2. Integrated remote monitoring technology/devices, e.g. smart scales, activity tracking devices.
3. Individualized weight management and exercise recommendations based on data collected from web/mobile app/devices to be delivered via web/mobile app/Smartphone; participants will not travel to a clinical facility for the intervention.

The objectives are:

1. to further develop the H.E.A.L.T.H. intervention by merging components of the H.E.A.L.T.H. program, remote monitoring technology components, e.g. activity tracking devices, smart scales, and direct/individualized weight management and exercise feedback into a single and comprehensive intervention that targets weight and fat loss, improved fitness, improved sleep, and personal well-being for Soldiers and their family members.
2. Compare body weight, body fat, and activity changes associated with participation in the H.E.A.L.T.H Intensive intervention for six months and a six-month website only phase/follow-up phase, in comparison to participation in a wait-list control group; and
3. Evaluate blood biomarkers associated with changes in body weight. Evaluate changes in gut bacteria associated with body weight.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female Soldiers who are members of the Louisiana National Guard

   * Direct family member of the LANG member who is enrolled in the study and will participate with the Soldier
2. ≥18 years old
3. For Soldiers: BMI ≥ 25, AND who exceeds Screening Table Weight AND maximum allowed body fat as outlined by AR600-9 Army regulations For Family Member: BMI ≥ 25
4. Has no known deployments (to the best of their knowledge) for one year upon beginning the study

Exclusion Criteria:

1. Soldiers and family members younger than 18 years of age
2. Soldiers and family members who are pregnant
3. Soldiers and family members who cannot read
4. Soldiers and family members who do not have daily access to wifi
5. Soldiers and family members who do not have access to a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Weight at 6 Months and 12 Months | Baseline, 6 Months, 12 Months
  Standard Weight Scale

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Stewart, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No